CLINICAL TRIAL: NCT02968940
Title: A Phase II, Open-label, Single Arm, Multicenter Study of Avelumab With Hypofractionated Radiation in Adult Subjects With Transformed IDH Mutant Glioblastoma
Brief Title: Avelumab With Hypofractionated Radiation Therapy in Adults With Isocitrate Dehydrogenase (IDH) Mutant Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01179
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Glioblastoma
Keywords: Programmed cell death protein 1 (PD-1); Programmed death-ligand 1 (PD-L1); Immunotherapy; Hypofractionated Radiotherapy (HFRT); Isocitrate dehydrogenase (IDH); Glioma
MeSH Terms: conditions — Glioblastoma; Parkinson Disease 4, Autosomal Dominant Lewy Body; Glioma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab and hypofractionated radiation therapy(HFRT) (Experimental): * Avelumab 10 mg/kg intravenously (IV) every 2 weeks.
  * Hypofractionated radiation therapy to a total dose of 30 Gy, delivered in 6 Gy per fraction for 5 consecutive daily fractions
  Interventions: Biological: Avelumab; Radiation: Hypofractionated radiation therapy (HFRT)

INTERVENTIONS:
Biological: Avelumab — Avelumab 10 mg/kg intravenously (IV) every 2 weeks
  Other Names: MSB0010718C
Radiation: Hypofractionated radiation therapy (HFRT) — Hypofractionated radiation therapy to a total dose of 30 Gy, delivered in 6 Gy per fraction for 5 consecutive daily fractions

SUMMARY:
The purpose of this study is to test how safe and effective treatment with the combination of Avelumab and radiation is for IDH mutant gliomas that have transformed to glioblastoma after chemotherapy.

DETAILED DESCRIPTION:
The active pharmaceutical ingredient in Avelumab (MSB0010718C) is a fully human antibody of the immunoglobulin gamma-1 (IgG1) isotype that specifically targets and blocks the Programmed death-ligand 1(PD-L1) for Programmed cell death protein 1 (PD-1).

Avelumab binds PD-L1 and blocks the interaction between PD-L1 and PD-1. This removes the suppressive effects of PD-L1 on anti-tumor cluster of differentiation 8 (CD8)+ T cells, resulting in the restoration of cytotoxic T cell response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years.
2. Documentation of IDH1 or IDH2 mutation in any tumor specimen.
3. Pathologic evidence (either diagnostic pathology slides or pathology report) of a diagnosis of WHO grade II or III glioma prior to treatment with temozolomide or PCV chemotherapy.
4. Histopathological evidence of glioblastoma (WHO grade IV) on a progressive tumor specimen after treatment with temozolomide or PCV chemotherapy. The diagnosis of glioblastoma must be confirmed on central review by a study-designated neuropathologist at NYULMC at screening.

Exceptions to this eligibility include the following:

a. Any progressive glioma with IDH1 or IDH2 mutation, regardless of WHO grade, histopathological diagnosis, or prior therapy, will be eligible if the progressive tumor specimen is found to have one of the genetic alterations below:

1. ≥20 somatic mutations per Mb by whole-exome sequencing
2. High mutation burden or microsatellite instability (MSI) identified by Foundation Medicine panel next-generation sequencing (FoundationOne®, FoundationOne CDx™). Foundation Medicine's threshold for high mutation burden (HMB) in their panel NGS assays is ≥20 somatic mutations per Mb. Foundation Medicine's panel NGS assay has been validated by whole-exome and whole-genome sequencing to correlate tightly with tumor mutation burden (R2 = 0.94).96
3. Mutation in a mismatch repair gene or other genes known to be associated with hypermutator phenotypes or microsatellite instability, including but not limited to MSH2, MSH6, MLH1, POLE, PMS2, POLD as determined by validated methods.
4. Microsatellite instability as identified by polymerase chain reaction (PCR) or other validated methods.

   b. Progressive oligodendroglioma (with 1p/19q codeletion) that has hallmark histopathological features of glioblastoma (i.e. necrosis, pseudopalisading necrosis, or microvascular proliferation) is eligible as IDH1/2 mutant, 1p/19q codeleted oligodendrogliomas that have progressed after chemotherapy have been shown to develop hypermutation phenotype.
5. Availability of a paraffin-embedded or frozen tumor-tissue block with a minimum of 1 cm2 of tumor surface area from a tissue specimen that demonstrates pathological transformation to glioblastoma (WHO grade IV) or a progressive specimen that harbors one of the genetic alterations specified in Inclusion Criteria 4a. a. If a tumor block cannot be submitted, then 20 unstained slides (preferably 10 slides from two different tumor blocks from the same surgery) from the tumor specimen must be submitted.
6. Patients must have had treatment with temozolomide, lomustine (CCNU) or PCV [procarbazine, lomustine (CCNU), vincristine] chemotherapy prior to histopathologic transformation to glioblastoma or prior to identification of one of the genetic alterations specified in Inclusion

Criteria 4a. Notes or records from the treating oncologist are required for documentation of treatment history. Prior treatment with at least one of the following chemotherapy schedules is required to be eligible:

1. At least one 6 week course of continuous daily temozolomide
2. At least six 28-day cycles given in one of the following schedules:

   1. Daily for 5 days of a 28-day cycle
   2. Daily for 21 days of a 28-day cycle
   3. Daily for 14 days of a 28-day cycle
   4. Alternating 7 days on/7 days per 28-day cycle
   5. Continuous daily dosing of a 28-day cycle.
3. Other schedules of temozolomide may be considered after discussion with the overall Principal Investigator.
4. At least 3 cycles of PCV or lomustine (CCNU) chemotherapy. 7. Patients who received anti-tumor therapy after histopathologic transformation to glioblastoma must have shown unequivocal radiographic evidence of tumor progression by contrast-enhanced MRI scan (or CT scan if MRI is contraindicated).

   8. Patients must have had prior CNS radiotherapy for their glioma, including standard doses for lowgrade or high-grade glioma as well as non-standard dose and fractionation, including hypofractionated regimens, stereotactic radiosurgery, etc.

   9. Patients can have had any number of prior therapies, including but not limited to molecularly targeted therapies and anti-angiogenic therapies, however they must have had prior chemotherapy with either temozolomide or lomustine as per Eligibility Criteria 6.

   10. Karnofsky performance status of ≥60. 11. Interval of at least 6 months from the completion of any prior radiotherapy and registration. If patients have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

a. New areas of tumor outside the original radiotherapy fields as determined by the investigator, or b. Histologic confirmation of tumor through biopsy or resection, or c. Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than pseudoprogression or radiation necrosis obtained within 28 days of registration AND an interval of at least 90 days between completion of radiotherapy and registration.

12. The following time periods must have elapsed prior to start of study treatment, the following time periods must have elapsed:

1. 5 half-lives from any investigational agent
2. 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas)
3. 6 weeks from antibodies
4. Prior treatment with other immune modulating agents within fewer than 4 weeks prior to the first dose of Avelumab. 1. Examples of immune modulating agents include blockers of CTLA-4, 4-1BB (CD137), OX-40, therapeutic vaccines, or cytokine treatments.
5. 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.

   13. An interval of at least 2 weeks (to start of study agent) between prior surgical resection or one week for stereotactic biopsy.

   14. Adequate hematologic, hepatic, and renal function defined by absolute neutrophil count ≥1.5 x 109/L, hemoglobin >9 g/dL, platelet count ≥ 100 x 109/L (may have been transfused), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN), total bilirubin ≤1.5 x ULN, and estimated creatinine clearance (CrCl) ≥ 30 mL/min according to the Cockcroft-Gault formula or local institutional standard method.

   15. Women of child-bearing potential (WOCBP) and men able to father a child must agree to use highly effective contraception while on study drug and for 30 days after the last dose of Avelumab. WOCBP must have a negative pregnancy test within 28 days of initiation of dosing.

Highly effective contraceptive measures include: stable use of oral contraceptives such as combined estrogen and progestogen and progestogen only hormonal contraception or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; intrauterine hormone-releasing system (IUS); bilateral tubal ligation; vasectomy and sexual abstinence.

1. Contraception is not required for men with documented vasectomy.
2. Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential.
3. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

   16. Willing to and capable of providing written informed consent prior to any study related procedures.

   17. Ability and willingness to comply with all study requirements, including scheduled visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Investigational drug use within 28 days of the first dose of Avelumab.
2. Planned participation in another study of an investigational agent or investigational device or use of a therapeutic device intended for therapy of glioma.
3. Prior therapy with an agent that blocks the PD-1/PD-L1 pathway.
4. Primary brainstem or spinal cord tumor.
5. Diffuse leptomeningeal disease at recurrence
6. Recurrent infratentorial tumor
7. Prior re-irradiation or stereotactic radiosurgery for recurrent disease at the same tumor location intended for HFRT in this study.
8. Maximal tumor diameter >4 cm
9. Patients with evidence of significant intracranial mass effect that requires >4 mg of dexamethasone or bioequivalent per day for 5 consecutive days for management of symptoms at any time within 14 days of registration.

   1. Subjects on a standard high-dose steroid taper after craniotomy may receive a higher dose of corticosteroids within 14 days of registration, however must be at a dose ≤4 mg of dexamethasone or bioequivalent per day within 5 days prior to registration.
   2. Administration of steroids through a route known to result in a minimal systemic exposure [i.e., intranasal, intraocular, inhaled, topical, or local injection (e.g., intra-articular injection) corticosteroids (<5% of body surface area)] are permitted.
   3. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are at doses ≤ 10 mg prednisone or bioequivalent per day.
   4. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are allowed.
10. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. The following are not exclusions:

    a. Patients with diabetes type I, vitiligo, hypo- or hyperthyroid diseases, or psoriasis not requiring systemic immunosuppressive treatment are eligible.
11. Prior organ transplantation, including allogeneic stem cell transplantation.
12. Known history of, or any evidence of active, non-infectious pneumonitis within the last 5 years.
13. Known prior, severe hypersensitivity (NCI-CTCAE v4.03 Grade 3 or 4) to investigational product or any component in its formulations including known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
14. Active infection requiring systemic therapy.
15. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
16. Positive test for Hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus (HCV antibody) at screening indicating acute or chronic infection.
17. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
18. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
19. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment, are acceptable.
20. Patients with another active cancer [excluding basal cell carcinoma, cervical carcinoma in situ or melanoma in situ]. Prior history of other cancer is allowed, as long as there was no active disease within the prior 2 years.
21. Pregnant or breastfeeding (negative serum or urine pregnancy test required for women of childbearing potential), or unable to maintain use of contraception while on study and for 30 days after the last dose of Avelumab.
22. Known alcohol or drug abuse
23. All other unstable, severe, or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
24. Any condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Kurz, MD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (4):
- United States (4):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Laura & Isaac Perlmutter Cancer Center & NYU Langone Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Avelumab and Hypofractionated Radiation Therapy(HFRT): * Avelumab 10 mg/kg intravenously (IV) every 2 weeks.
  * Hypofractionated radiation therapy to a total dose of 30 Gy, delivered in 6 Gy per fraction for 5 consecutive daily fractions
  Avelumab: Avelumab 10 mg/kg intravenously (IV) every 2 weeks
  Hypofractionated radiation therapy (HFRT): Hypofractionated radiation therapy to a total dose of 30 Gy, delivered in 6 Gy per fraction for 5 consecutive daily fractions
Period: Overall Study
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 45 [31.5 to 54.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities
Description: Subjects are evaluable for DLTs (defined in section 5.2.1.2) if they have received at least one dose of Avelumab, have completed HFRT per protocol and have completed safety assessments over the entire DLT evaluation period (days 1 through 28).
Time Frame: Day 28
Measure: Number; unit: Events meeting DLT Criteria
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
Number analyzed (Participants) | 6
Events meeting DLT Criteria | 0

2. Primary Outcome: Median Progression-free Survival (PFS6)
Description: PFS, defined as the time between treatment initiation and first occurrence of disease progression or death, will be censored at last follow-up if the patient remained alive without disease progression
Time Frame: Month 6
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
Number analyzed (Participants) | 6
Months | 4.2 [1.4 to 5.7]

3. Secondary Outcome: Median Overall Survival (OS)
Description: OS will be determined from the time of treatment initiation until the time of death, with OS being censored at last follow-up if the patient remained alive
Time Frame: Month 12
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
Number analyzed (Participants) | 6
Months | 10.1 [6.8 to 12]

4. Secondary Outcome: Median Progression-free Survival (PFS12)
Description: as for outcome 2
Time Frame: Month 12
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
Number analyzed (Participants) | 6
Months | 4.2 [1.4 to 5.7]

ADVERSE EVENTS:
Time Frame: 12 months
Description: regular investigator assessment
Arm/Group | Avelumab and Hypofractionated Radiation Therapy(HFRT)
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab and Hypofractionated Radiation Therapy(HFRT) (N=6)
Edema cerebral (Nervous system disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Infusion related reaction (General disorders) | 1
Other, radiation vasculopathy (Vascular disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab and Hypofractionated Radiation Therapy(HFRT) (N=6)
White blood cell decreased (Investigations) | 4
Vomiting (Gastrointestinal disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Spasticity (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Sun burn (Skin and subcutaneous tissue disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinus pain (Nervous system disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Seizure (Nervous system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Pyramidal tract syndrome (Nervous system disorders) | 2
Psychosis (Psychiatric disorders) | 1
Platelet count decreased (Investigations) | 2
Pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Paresthesia (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Memory impairment (Nervous system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypotension (Vascular disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Headache (Nervous system disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Tongue sores (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Facial nerve disorder (Nervous system disorders) | 1
Edema limbs (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Creatinine increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Concentration impairment (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Chills (General disorders) | 1
CD4 lymphocytes decreased (Investigations) | 3
Blurred vision (Eye disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Anxiety (Psychiatric disorders) | 2
Anorectal infection (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Abdominal Pain (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02968940/Prot_SAP_000.pdf